CLINICAL TRIAL: NCT02114021
Title: Effect of Betamethasone Gel and Lidocaine Jelly Applied Over Tracheal Tube Cuff on Post Operative Sore Throat, Cough and Hoarseness of Voice on the Patients
Brief Title: Effect of Betamethasone Gel and Lidocaine Jelly on Sore Throat, Cough and Hoarseness of
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Fatemeh Shahbazi, Principal Investigator, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08/13/1019
Record Dates: First submitted 2014-04-07; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Sore Throat; Cough
Keywords: Syndrome incidence after intubation; Betamethasone gel; lidocaine jelly; sore throat; cough; hoarseness of voice
MeSH Terms: conditions — Pharyngitis; Cough; Hoarseness | interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- betamethasone gel (Experimental): betamethasone gel (over tracheal tube cuff) compared with distilled water on the post intubation syndrome incidence.
  Interventions: Drug: betamethasone gel; Drug: distilled water
- lidocaine jelly (Experimental): lidocaine jelly (over tracheal tube cuff) compared with distilled water on the post intubation syndrome incidence.
  Interventions: Drug: lidocaine jelly; Drug: distilled water
- distilled water (Placebo Comparator): betamethasone gel and lidocaine jelly (over tracheal tube cuff) compared with distilled water on the post intubation syndrome incidence.

INTERVENTIONS:
Drug: betamethasone gel — betamethasone gel (over tracheal tube cuff) compared with distilled water on the post intubation syndrome incidence.
  Arms: betamethasone gel
Drug: lidocaine jelly — the effect of lidocaine jelly (over tracheal tube cuff) compared with distilled water on the post intubation syndrome incidence.
  Arms: lidocaine jelly
Drug: distilled water — The effect of betamethasone gel and lidocaine jelly (over tracheal tube cuff) compared with distilled water on the post intubation syndrome incidence.
  Arms: betamethasone gel; lidocaine jelly

SUMMARY:
ABSTRACT:

The aim of this study was to investigate the effect of betamethasone gel and lidocaine jelly (over tracheal tube cuff) compared with distilled water on the post intubation syndrome incidence. This study has not been carried out in Iran.

99 patients of either sex undergoing elective surgery were recruited in a single blind randomized study. The patients, using randomization table, were divided into three groups. Anesthetics and medications used during surgery were similar for all the patients.

For the all patients, the incidence of postoperative sore throat, cough and hoarseness of the voice in the different follow-up periods (1, 6 and 24 hours) based on the different types of medications were obtained.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years<age>15 years
2. no acute upper respiratory infections and no sore throat
3. candidate for elective surgery unrelated to the throat
4. The lack of airways difficulties
5. candidate for general anesthesia with intubation
6. no contraindications for receiving steroid
7. surgery time < 240 minutes
8. intubation up to 2 times
9. tracheal tube cuff pressure = 25-30 cm H2o
10. fasting for 8-6 hours prior to surgery
11. ASA I and ASAII and
12. Surgery under general anesthesia and endotracheal intubation

Exclusion Criteria:

1. use of nasogastric tube or throat packs
2. patients with upper respiratory tract infection
3. patients on steroid therapy were excluded from the study

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
sore throat | 24 hours after surgery
  For the all the patients, the incidence of postoperative cough in 24 hours follow-up based on the different types of medications were obtained (using questionnaire).
cough | 1 hour after surgery
  For the all the patients, the incidence of postoperative cough in 1 hour follow-up periods based on the different types of medications were obtained (using questionnaire).
hoarseness of voice | 1 hour after surgery
  For the all patients, the incidence of postoperative hoarseness of the voice in 1 hour follow-up period based on the different types of medications were obtained (using questionnaire).
sore throat | 1 hour after surgery
  For the all the patients, the incidence of postoperative cough in 1 hour follow up based on the different types of medications were obtained (using questionnaire).
sore throat | 6 hours after surgery
  For the all the patients, the incidence of postoperative cough in 6 hours follow-up based on the different types of medications were obtained (using questionnaire).
cough | 6 hours after surgery
  For the all the patients, the incidence of postoperative cough in 6 hours follow-up periods based on the different types of medications were obtained (using questionnaire).
cough | 24 hours after surgery
  For the all the patients, the incidence of postoperative cough in 24 hours follow-up periods based on the different types of medications were obtained (using questionnaire).
hoarseness of voice | 6 hours after surgery
  For the all patients, the incidence of postoperative hoarseness of the voice in 6 hours follow-up period based on the different types of medications were obtained (using questionnaire).
hoarseness of voice | 24 hours after surgery
  For the all patients, the incidence of postoperative hoarseness of the voice in 24 hours follow-up period based on the different types of medications were obtained (using questionnaire).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Booali Hospital, Islamic Azad University,, Tehran, Iran